CLINICAL TRIAL: NCT00435266
Title: The Effect of Remote Preconditioning in Primary Percutaneous Intervention of Acute ST Elevation Myocardial Infarction
Brief Title: Remote Ischemic Preconditioning in Primary PCI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Falck, Denmark (Unknown); Doctor's ambulance Services, Aarhus, Denmark (Unknown); Royal Brompton & Harefield NHS Foundation Trust (Other); The Hospital for Sick Children (Other)
Responsible Party: Hans Erik Bøtker, MD. Ph.D., Professor, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 95093546-1
Record Dates: First submitted 2007-02-13; First posted 2007-02-14 (Estimated); Last update posted 2009-02-17 (Estimated); Status verified 2009-02

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; remote; preconditioning; perconditioning; cardioprotection
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Remote ischemic preconditioning
  Interventions: Procedure: Remote ischemic preconditioning
- 2 (No Intervention)
  Interventions: Procedure: Remote ischemic preconditioning

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — Inflation of blood pressure cuff 4 x 5 minutes during transportation to primary PCI

SUMMARY:
Primary percutaneous coronary intervention (pPCI) is the preferred treatment in ST elevation myocardial infarction (STEMI). The infarct-related artery (IRA) can be opened in more than 90% of the patients. However, STEMI patients still end up with a persistent perfusion defect of highly variable magnitude indicating that adjunctive treatment may add further protection against tissue damage. Ischemic preconditioning (IPC) is an intervention by which myocardium threatened by ischemia is exposed to short and repeated sublethal ischemic episodes prior to sustained ischemia (local IPC). A systemic response with protection of more remote organs (remote IPC (rIPC)) also can be induced. We have recently found that the infarct reducing effect can be obtained by obstruction of an extremity even though the remote stimulus is initiated during sustained occlusion of a coronary artery, the so-called remote preconditioning (rPerC). The clinical perspective is now to examine if rPerC can reduce the infarct size in patients with unpredictable ischemia in ST elevation myocardial infarction (STEMI). We perform a randomized study where patients en route for pPCI are allocated to either rPerC or a standard treatment to evaluate whether the tissue damage can be reduced. Effect measure will be infarct size determined by scintigraphy (final infarct size and salvage).

DETAILED DESCRIPTION:
Primary percutaneous coronary intervention (pPCI) is the preferred treatment in ST elevation myocardial infarction (STEMI). The infarct-related artery (IRA) can be opened in more than 90% of the patients. However, STEMI patients still end up with a persistent perfusion defect of highly variable magnitude indicating that adjunctive treatment may add further protection against tissue damage. Ischemic preconditioning (IPC) is an intervention by which myocardium threatened by ischemia is exposed to short and repeated sublethal ischemic episodes prior to sustained ischemia (local IPC). A systemic response with protection of more remote organs (remote IPC (rIPC)) also can be induced. We have recently found that the infarct reducing effect can be obtained by obstruction of an extremity even though the remote stimulus is initiated after sustained occlusion of a coronary artery, the so-called remote preconditioning (rPerC). The clinical perspective is now to examine if rPerC can reduce the infarct size in patients with unpredictable ischemia in ST elevation myocardial infarction (STEMI). We perform a randomized study where patients en route for pPCI are allocated to either rPerC or a standard treatment to evaluate whether the tissue damage can be reduced. Effect measure will be infarct size determined by scintigraphy (final infarct size and salvage).

Purpose

The purpose of the present study is to examine the utility of rPerC in STEMI patients treated with pPCI. The effect will be evaluated by 1) limitation of infarct size (salvage and final infarct size) determined by myocardial scintigraphy (SPECT), 2) electrocardiographic and angiographic signs of tissue perfusion, 3) release of ischemic markers 5) echocardiographic markers of left ventricular function and 5) clinical end-points (Major Adverse Cardiac Events (MACE: death, reinfarction, need for revascularisation, invalidating stroke)) at discharge and after 30 days.

Description and evaluation of the ethical aspects of the study

Study patients treated with pPCI are randomized to pretreatment with rPerC or no pretreatment (control group). The randomization will take place in the ambulance or at the local hospital. With the aim of not causing unnecessary delays, the pretreatment is discontinued if the patient arrives at the cath. lab. before the pretreatment is completed.The discomfort in connection with the pretreatment has been shown to be minimal.

Information regarding study population

The patients are recruited among patients admitted or transferred to Department of Cardiology B, Skejby Sygehus for pPCI treatment for STEMI.

Review on the methods used

rPerC The pretreatment in the rPerC group comprises 4 x (5 min. occlusion of right upper extremity followed by 5 min. reperfusion) which is performed during the transportation towards Skejby Sygehus. The occlusion is obtained by inflation of a blood pressure tourniquet placed on the patient's right thigh to 200 mm Hg or 25 mmHg above the patient's systolic blood pressure when higher than 200 mm Hg.

Angiography The initial angiography is performed in at least two planes after administration of nitroglycerin 0.2 mg intracoronary and filmed at 25 frames/sec. The lesion should be placed centrally in the picture with the tip of the guiding catheter visual in the picture.

The final angiography is performed in the same planes as the initial angiography and after administration of nitroglycerin 0.2 mg intracoronary. The angiography is filmed at 25 frames/sec. and the filming is continued until a clear projection of sinus coronarius. The angiogram is filmed with and without magnification with the aim of projecting the periphery of the vessels.

The final angiography is performed two minutes after the last dilatation - provided that the patient is hemodynamically stable.

Percutaneous intervention and antithrombotic treatment The patients will have PCI performed in accordance with the existing procedures and guidelines at Skejby Hospital.

Electrocardiogram (ECG) and monitoring Continuous 12-lead ST-monitoring is initiated on scene by use of a commercial monitor-defibrillator (LIFEPAK 12, Medtronic Emergency Response Systems, USA), and continued during transport to the local hospital (if not bypassed) and during transfer to the interventional hospital. On arrival at the interventional hospital traditional ECG electrodes are replaced by radiolucent carbon fiber lead wire electrodes (Ambu Blue Sensor QR electrodes, Ambu A/S, Denmark) enabling ST-monitoring to be continued during and 90 minutes following PCI. The analog ECG signals sampled by the system are digitized at a sample rate of 500 Hz for processing by the GE/Marquette Medical Systems 12SL ECG interpretive algorithm. At 30-second interval the ST-monitoring program generates a median QRST-complex for all 12 leads based on a 10-second epoch of ECG data. From each of these median QRST-complexes the program estimates the ST-deviation at the STM point, halfway between the J-point of the QRS complex and the start of the T-wave. If a 0.1 mV change in ST-deviation lasts for 2.5 minutes then the software automatically acquires and stores a 10-second 12-lead ECG waveform. All 12-lead ECG waveforms and continuous ST-monitoring data are transferred to a personal computer and stored by a random key for subsequent blinded analysis at the Core Lab. at Skejby Sygehus.

Biochemical ischemia markers Circulating concentrations of troponin T (TnT) is measured at arrival, 8-12 hours, 20-24 hours and finally 90-102 hours after symptom onset.

Scintigraphic methods Two scintigraphic examinations are performed to determination of area at risk (AAR), final infarct size (FIS), regional wall motion and regional wall thickening respectively.

Area at risk (AAR): (That part of left ventricle that is without perfusion prior to PCI) Determined by tracer injection during ongoing coronary occlusion which means tracer injection prior to PCI but imaging after pPCI.

Final infarct size (FIS): (That part of left ventricle that is without perfusion 1 month after PCI) Determined by myocardial scintigraphy at rest 1 month after pPCI.

The following parameters are calculated:

Salvage : AAR minus FIS (% of left ventricle) Salvage index (%): Salvage / AAR. Left ventricular ejection fraction (LVEF) (%): (EDV - ESV)/EDV. Each myocardial scintigraphy is performed after administration of 700 ± 10% MBq 99mTc-Sestamibi as an intravenous bolus injection. Acquisition is performed as gated SPECT within 8 hours after tracer injection. The myocardial perfusion is analyzed and quantitized by the use of the interpretation software QPS and QGS. At each examination partly myocardial perfusion defect as a percentage of left ventricular myocardium, partly left ventricular end-diastolic and end-systolic volume (EDV and ESV) and partly regional wall motion and wall thickening is determined.

Design and data registration The patients are randomized to pPCI treatment with or without prior rIPC. All data analyzes from the study will be analyzed blinded regarding to the patient's randomization.

For each participant included in the study, a case record form (CRF) is filled in.

Definition and characteristic of effect parameters and other registered data A consecutive patient registration is performed by a characteristic of the study population and a registration of causes of exclusion. Clinical, angiographic and procedure related variables as in the West-Danish Heart Database will be used.

Data evaluation For each of the primary and secondary clinical effect parameters, a comparative examination of the rPerC and not rPerC treated patient groups is performed.

Statistics Dimensioning the study: Previous investigations have shown that area at risk in connection with STEMI is approximately 30% of left ventricle. Experiences from investigations at Department of Cardiology B and Department of Nuclear Medicine, Skejby Sygehus, have shown that the final infarct size in STEMI patients treated with pPCI is approximately 15%.

It is estimated that a 20% reduction in infarct size (e.g. from 15% to 12%) will be clinically relevant. With a spreading of the infarct size of 15%, which are in accordance with our previous findings, detection of such a reduction with a risk of type 2 errors of 80% (2α=0.80) will require 109 patients in each group. We plan inclusion of a total of 250 patients to secure complete data.

The study will be analyzed after intention-to-treat principles. A final specification will be performed with unpaired parametric or non parametric statistics.

ELIGIBILITY:
Inclusion Criteria:

1. Acute chest pain or equivalent symptoms during > 30 minutes.
2. Duration of symptoms < 12 hours.
3. Cumulated ST elevation > 2 mm in two contiguous leads.
4. Age ≥ 18 years.
5. Informed consent

Exclusion Criteria:

1. Previous by-pass surgery.
2. Pulseless femoral artery.
3. Left bundle branch block in ECG (LBBB).
4. Acute MI and/or treatment with thrombolysis within 30 days.
5. Patients treated with cooling or patients who have had cardiac arrest.
6. Diabetic patients
7. Patients with arteriovenous shunts for the purpose of hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Salvage index (% of left ventricle): Salvage / Area at Risk (AAR) by SPECT | 30 days

SECONDARY OUTCOMES:
Final infarct size. | 30 days
Proportion of patients achieving ≥70% ST-resolution 90 minutes following pPCI | 90 minutes
Proportion of patients achieving spontaneous ST-resolution before pPCI | Immediate
Proportion of patients with increase in ST-elevation during pPCI. | Immediate
Time from first ECG to ≥70% ST-resolution (continuous parameter) | Minutes
Time from first wire to ≥70% ST-resolution (continuous parameter) | Minutes
ST resolution immediately after ending the procedure (evaluated in relation to ST elevation on ECG obtained just prior to the pPCI procedure). | Minutes
Prompt angiographic success: | Immediate
Corrected TIMI frame count (cTFC). | Minutes
TIMI flow measured immediately after ending the interventional procedure. | Minutes
Myocardial blush. | Minutes
Procedure duration. | Minutes
Total duration of hospitalisation. | Days
MACE after 30 days. | 30 days
TnT release - determined 90-102 hours after symptom onset. | 90-102 hours
Echocardiographic data (acute and after 1 month): | 30 days
WMI. | 30 days
Left ventricular ejection fraction (LVEF) (%): (EDV - ESV)/EDV. | 30 days
Myocardial scintigraphy data: | 30 days
Regional wall motion and regional thickening. | 30 days
Technical success. | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Torsten T Nielsem, MD, Study Director — Aarhus University Hospital; Hans Erik Bøtker, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Cardiology, Aarhus University Hospital Skejby, Aarhus N, Denmark

REFERENCES:
- [Result] Schmidt MR, Smerup M, Konstantinov IE, Shimizu M, Li J, Cheung M, White PA, Kristiansen SB, Sorensen K, Dzavik V, Redington AN, Kharbanda RK. Intermittent peripheral tissue ischemia during coronary ischemia reduces myocardial infarction through a KATP-dependent mechanism: first demonstration of remote ischemic perconditioning. Am J Physiol Heart Circ Physiol. 2007 Apr;292(4):H1883-90. doi: 10.1152/ajpheart.00617.2006. Epub 2006 Dec 15. PMID 17172279
- [Result] Kristiansen SB, Henning O, Kharbanda RK, Nielsen-Kudsk JE, Schmidt MR, Redington AN, Nielsen TT, Botker HE. Remote preconditioning reduces ischemic injury in the explanted heart by a KATP channel-dependent mechanism. Am J Physiol Heart Circ Physiol. 2005 Mar;288(3):H1252-6. doi: 10.1152/ajpheart.00207.2004. Epub 2004 Oct 21. PMID 15498829
- [Result] Kristiansen SB, Lofgren B, Stottrup NB, Khatir D, Nielsen-Kudsk JE, Nielsen TT, Botker HE, Flyvbjerg A. Ischaemic preconditioning does not protect the heart in obese and lean animal models of type 2 diabetes. Diabetologia. 2004 Oct;47(10):1716-21. doi: 10.1007/s00125-004-1514-4. Epub 2004 Oct 7. PMID 15480537
- [Result] Kharbanda RK, Mortensen UM, White PA, Kristiansen SB, Schmidt MR, Hoschtitzky JA, Vogel M, Sorensen K, Redington AN, MacAllister R. Transient limb ischemia induces remote ischemic preconditioning in vivo. Circulation. 2002 Dec 3;106(23):2881-3. doi: 10.1161/01.cir.0000043806.51912.9b. PMID 12460865
- [Result] Cheung MM, Kharbanda RK, Konstantinov IE, Shimizu M, Frndova H, Li J, Holtby HM, Cox PN, Smallhorn JF, Van Arsdell GS, Redington AN. Randomized controlled trial of the effects of remote ischemic preconditioning on children undergoing cardiac surgery: first clinical application in humans. J Am Coll Cardiol. 2006 Jun 6;47(11):2277-82. doi: 10.1016/j.jacc.2006.01.066. Epub 2006 May 15. PMID 16750696
- [Derived] Pryds K, Bottcher M, Sloth AD, Munk K, Rahbek Schmidt M, Botker HE; CONDI Investigators. Influence of preinfarction angina and coronary collateral blood flow on the efficacy of remote ischaemic conditioning in patients with ST segment elevation myocardial infarction: post hoc subgroup analysis of a randomised controlled trial. BMJ Open. 2016 Nov 24;6(11):e013314. doi: 10.1136/bmjopen-2016-013314. PMID 27884851
- [Derived] Pryds K, Terkelsen CJ, Sloth AD, Munk K, Nielsen SS, Schmidt MR, Botker HE; CONDI Investigators. Remote ischaemic conditioning and healthcare system delay in patients with ST-segment elevation myocardial infarction. Heart. 2016 Jul 1;102(13):1023-8. doi: 10.1136/heartjnl-2015-308980. Epub 2016 Feb 24. PMID 26911520
- [Derived] Sloth AD, Schmidt MR, Munk K, Schmidt M, Pedersen L, Sorensen HT, Botker HE; CONDI Investigators. Impact of cardiovascular risk factors and medication use on the efficacy of remote ischaemic conditioning: post hoc subgroup analysis of a randomised controlled trial. BMJ Open. 2015 Apr 2;5(4):e006923. doi: 10.1136/bmjopen-2014-006923. PMID 25838505
- [Derived] Botker HE, Kharbanda R, Schmidt MR, Bottcher M, Kaltoft AK, Terkelsen CJ, Munk K, Andersen NH, Hansen TM, Trautner S, Lassen JF, Christiansen EH, Krusell LR, Kristensen SD, Thuesen L, Nielsen SS, Rehling M, Sorensen HT, Redington AN, Nielsen TT. Remote ischaemic conditioning before hospital admission, as a complement to angioplasty, and effect on myocardial salvage in patients with acute myocardial infarction: a randomised trial. Lancet. 2010 Feb 27;375(9716):727-34. doi: 10.1016/S0140-6736(09)62001-8. PMID 20189026
- See also: Aarhus University webpage — http://www.au.dk/en